CLINICAL TRIAL: NCT00567476
Title: A Randomized, Open-label, Multicenter Study to Evaluate the Effect of Xolair (Omalizumab) as Add-on Therapy to Inhaled Corticosteroid + Long-Acting Beta Agonist in Fixed or Flexible Dosing Compared to Isolated Inhaled Corticosteroid + Long-Acting Beta Agonist in Fixed or Flexible Dosing in the Asthma-Related Quality of Life in Patients With Severe Persistent Allergic Asthma
Brief Title: Omalizumab Use and Asthma-Related Quality of Life in Patients With Severe Persistent Allergic Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIGE025ABR01
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Results first posted 2011-05-23 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Asthma
Keywords: Asthma, anti-immunoglobulin E, omalizumab
MeSH Terms: conditions — Asthma | interventions — Omalizumab; Albuterol; Terbutaline

ARMS (2):
- Omalizumab + Conventional Therapy (Active Comparator): Omalizumab was administered subcutaneously every 2 or 4 weeks over a period of 20 weeks to provide a dose of at least 0.016 mg/kg per UI/ml of immunoglobulin E (IgE). Doses (mg) and dosing frequency were determined by serum total IgE level (IU/mL) and body weight (kg). Also, participants continued using their current formulation of inhaled corticosteroid (ICS) and long-acting beta 2-adrenergic agonist (LABA). Home use of nebulized beta 2-agonist was allowed for the treatment of symptoms of intercurrent bronchospasm or during an asthma exacerbation if this treatment regimen was already established prior to screening visit.
  Interventions: Drug: Omalizumab; Drug: Inhaled corticosteroids (ICS); Drug: Long-acting beta 2-adrenergic agonist (LABA); Drug: Short-acting beta 2-adrenergic agonist (SABA)
- Conventional Therapy (Active Comparator): Participants continued using their current formulation of inhaled corticosteroid (ICS) and a long-acting beta 2-adrenergic agonist (LABA). Home use of nebulized beta 2-agonist was allowed for the treatment of symptoms of intercurrent bronchospasm or during an asthma exacerbation if this treatment regimen was already established prior to screening visit.
  Interventions: Drug: Inhaled corticosteroids (ICS); Drug: Long-acting beta 2-adrenergic agonist (LABA); Drug: Short-acting beta 2-adrenergic agonist (SABA)

INTERVENTIONS:
Drug: Omalizumab — Omalizumab 150 to 375 mg was administered subcutaneously every 2 or 4 weeks to provide a dose of at least 0.016 mg/kg per UI/ml of IgE.
  Other Names: Xolair
  Arms: Omalizumab + Conventional Therapy
Drug: Inhaled corticosteroids (ICS) — Any ICS with proprietary drug and device > 500 mcg of fluticasone or equivalent
Drug: Long-acting beta 2-adrenergic agonist (LABA) — Fixed dose of LABA as prescribed prior to study entry
Drug: Short-acting beta 2-adrenergic agonist (SABA) — Home use of nebulized Β2-agonist such as salbutamol 5 mg or terbutaline 10 mg for symptoms of intercurrent bronchospasm.
  Other Names: salbutamol; terbutaline

SUMMARY:
This study investigated asthma-related quality of life in Brazilian patients using omalizumab.

ELIGIBILITY:
Inclusion criteria:

* 12 to 75 years-old during screening visit.
* Body weight > 20 kg and < 150 kg.
* Daily or persistent asthma symptoms.
* Night symptoms at least once a week.
* Forced expiratory volume in 1 second (FEV1) > 40% and < 80% of predicted normal value and continuing asthma symptoms.
* FEV1 increased > 12% from baseline within 30 minutes of inhaled (up to 400 mcg) or nebulized (up to 5 mg) salbutamol.
* Subject taking more than 500 mcg/day of fluticasone or equivalent associated to a long-acting β2-agonist.
* Inhaled corticosteroid and long-acting beta-2 adrenergic agonist (LABA) doses that remained fixed during the last 12 weeks prior to screening.
* Medical history of at least two episodes of asthma exacerbation treated with systemic corticoid or at least one severe asthma exacerbation treated with systemic corticoid and hospitalization or emergency room visit in the last 12 months prior to screening.
* Positive skin prick test (diameter of wheal > 3mm) to at least one perennial aeroallergen (dust mite, cat/dog dander, cockroaches), to which the subject was likely to be exposed during the study.
* Subject capable to read and understand asthma related quality of life questionnaire (Juniper's questionnaire).

Exclusion criteria:

* Pregnant, nursing female subjects.
* Female subjects without current acceptable contraceptive method.
* Previous history of allergy or hypersensitivity to omalizumab.
* Subjects with prior treatment with omalizumab.
* Subjects with medical history of psychiatric disorder.
* Subject had been treated with systemic corticosteroid for any reason other than asthma.
* Subject took β2 antagonist medication in the last 3 months prior to screening visit.
* Subject took protocol prohibited medication prior to screening.
* Medical history of food or drug related severe anaphylactoid reactions.
* Medical history of antibiotics allergy. Patients were included if the antibiotics to which they were allergic to were to be avoided for the entire duration of the study.
* Asthma related to non-steroidal anti-inflammatory drug (NSAID).
* Treatment of exacerbation in the 4 weeks prior to randomization.
* Other active lung diseases.
* Medical history of others uncontrolled diseases 3 months prior randomization (eg, infections, coronary heart diseases and metabolic diseases).
* Any history of cancer.
* Abnormal electrocardiogram (ECG), laboratory exams (clinically significant abnormalities), and chest X-ray (CXR).
* Evidence or history of drug or alcohol abuse.
* Airway infection (eg, pneumonia, acute sinusitis) 4 weeks prior to screening visit.
* Smokers or smoking history of > 10 pack-years.
* Subject that had been treated with investigational drugs over the past 30 days or during the course of the trial.
* Subject had elevated IgE levels for reasons other than allergy.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigator Site, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab + Conventional Therapy | Conventional Therapy
Started | 78 | 38
Completed | 70 | 34
Not Completed | 8 | 4
Not completed — Adverse Event | 2 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 4 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Administrative issues | 1 | 0
Not completed — Medical Decision | 0 | 1
Not completed — Non-adherence to protocol | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab + Conventional Therapy | Conventional Therapy | Total
Number analyzed (Participants) | 78 | 38 | 116
Age, Customized [Number; unit: Participants]
  > 12 years and < 25 years | 4 (13.1) | 4 (12.8) | 8
  ≥ 25 and < 35 years | 15 | 3 | 18
  ≥ 35 and < 55 years | 42 | 23 | 65
  ≥ 55 and < 65 years | 12 | 4 | 16
  ≥ 65 and < 75 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 29 | 89
  Male | 18 | 9 | 27

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With an Increase of More Than 1.5 in AQLQ Overall Score at 20 Weeks
Description: The AQLQ was administered to all patients at Baseline, Week 12 and Week 20. The 32 questions in the AQLQ were divided into four domains; activity limitations, symptoms, emotional function, and environmental stimuli. Individual questions are equally weighted. The overall AQLQ score is the mean of the responses to each of the 32 questions and ranges from 1 to 7. A score 7.0 indicates that the patient has no impairments due to asthma and score 1.0 indicates severe impairment.
Time Frame: Baseline and Week 20
Population: Patients who took at least one dose of double-blind study drug and who had at least one post-baseline safety or efficacy assessment made up the intent-to treat (ITT) population. Last observation carried forward (LOCF) approach was used. Scores of completed AQLQ at Week 12 were used at Week 20 for dropped out patients or for missing values.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omalizumab + Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 77 | 36
Percentage of participants | 40.3 [30.0 to 51.4] | 2.8 [0.5 to 14.2]

2. Secondary Outcome: Percentage of Participants With an Increase of More Than 0.5 in AQLQ Overall Score at Week 20
Description: The AQLQ was administered to all patients at Baseline, Week 12 and Week 20. The 32 questions in the AQLQ were divided into four domains; activity limitations, symptoms, emotional function, and environmental stimuli. Individual questions are equally weighted. The overall AQLQ score is the mean of the responses to each of the 32 questions and ranges from 1 to 7. AQLQ of each domain is the mean of the responses to each of the questions within that domain. A score 7.0 indicates that the patient has no impairments due to asthma and score 1.0 indicates severe impairment.
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omalizumab + Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 77 | 36
Percentage of participants | 70.1 [59.2 to 79.2] | 22.2 [11.7 to 38.1]

3. Primary Outcome: The Mean Change From Baseline to Week 20 in the Overall Asthma Quality of Life Questionnaire (AQLQ)
Description: The AQLQ was administered to all patients at Baseline, Week 12 and Week 20. The 32 questions in the AQLQ were divided into four domains; activity limitations, symptoms, emotional function, and environmental stimuli. Individual questions are equally weighted. The overall AQLQ score is the mean of the responses to each of the 32 questions, and ranges from 1 to 7. A score 7.0 indicates that the patient has no impairments due to asthma and a score of 1.0 indicates severe impairment.
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Omalizumab + Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 78 | 38
Units on a scale
  Baseline (n=77, 37) | 3.1 (1.0) | 3.1 (1.1)
  At Week 20 (n=78, 36) | 4.4 (1.4) | 3.0 (1.1)
  Change from baseline to week 20 (n=77, 36) | 1.2 (0.1) | -0.1 (0.1)

4. Secondary Outcome: The Mean Change From Baseline to the End of Study in AQLQ Domain Score
Description: AQLQ was administered to all patients at Baseline, Week 12 and Week 20, and prior to any clinic visit evaluation and drug administration.
  The 32 questions in the AQLQ were divided into four domains: activity limitations, symptoms, emotional function, and environmental stimuli. AQLQ domain scores were calculated by adding the responses to each of the questions in the domain and dividing by the number of questions in the domain. Each domain score was between 1 and 7. Score 7.0 meant that the patient had no impairments due to asthma and score 1.0 indicated severe impairment.
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Omalizumab + Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 78 | 38
Units on a scale
  Activity limitation score | 1.3 (0.1) | -0.2 (0.1)
  Symptoms score | 1.2 (0.2) | -0.2 (0.2)
  Emotional function score | 1.3 (0.2) | 0.0 (0.1)
  Environmental stimuli score | 1.2 (0.2) | 0.0 (0.2)

5. Secondary Outcome: Number of Asthma Exacerbation Episodes Per Participant
Description: For the purpose of evaluating efficacy, a clinically significant asthma exacerbation was defined as a worsening of asthma symptoms as judged clinically by the investigator, requiring doubling the baseline ICS dose for at least 3 days and/or treatment with rescue systemic (oral or IV) corticosteroids. The initiation of the above corticosteroid regimens marked the start of an asthma exacerbation episode and cessation of the additional corticosteroid regimens marked the end of an exacerbation episode.
Time Frame: From Baseline through 20 weeks
Population: All randomized patients who took at least one dose of double-blind study medication and who had at least one post-baseline safety or efficacy assessment made up the ITT population.
Measure: Number; unit: Participants
Arm/Group | Omalizumab + Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 78 | 38
Participants
  Patients with 1 episode | 25 | 12
  Patients with 2 episodes | 5 | 6
  Patients with 3 episodes | 3 | 1
  Patients with 4 episodes | 1 | 1
  Total number of patients with episodes | 34 | 20

6. Secondary Outcome: Percentage of Participants Using Rescue Medication
Description: When necessary, patients were allowed to take rescue medication using inhaled salbutamol or terbutaline for symptoms of intercurrent bronchospasm.
Time Frame: From Baseline through 20 Weeks
Population: All randomized patients who took at least one dose of double-blind study medication and who had at least one post-baseline safety or efficacy assessment made up the intention-to-treat (ITT) population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omalizumab + Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 78 | 38
Percentage of participants | 43.6 [33.1 to 54.6] | 44.7 [30.1 to 60.3]

7. Secondary Outcome: Free Days With no Rescue Medication
Description: When necessary, patients were allowed to take rescue medication using inhaled salbutamol or terbutaline for symptoms of intercurrent bronchospasm. Days with no rescue medication intake were the variable of interest for this analysis.
Time Frame: From Baseline through 20 weeks (140 days)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Omalizumab + Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 78 | 38
Days | 73.5 (39.4) | 74.9 (35.4)

8. Secondary Outcome: Mean Number of Puffs of Rescue Medication Taken Per Day
Description: When necessary, patients were allowed to take rescue medication using inhaled salbutamol or terbutaline for symptoms of intercurrent bronchospasm. The number of puffs taken during each 24 hour period was recorded in the patient dairy. The total number of puffs over 20 weeks of treatment was divided by the number of treatment days (140 days) to calculate the mean number of puffs per day.
Time Frame: From Baseline through 20 Weeks
Population: All randomized patients who took at least one dose of double-blind study medication and who had at least one post-baseline safety or efficacy assessment made up the intention-to-treat (ITT) population. Number of patients analyzed includes only those patients requiring rescue medication during the study.
Measure: Mean (Standard Deviation); unit: Puffs
Arm/Group | Omalizumab + Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 34 | 17
Puffs | 5.5 (4.1) | 6.4 (4.7)

9. Secondary Outcome: Physician's Global Assessment of Treatment Effectiveness
Description: At the end of Week 20 a global evaluation of the treatment effectiveness was performed by the investigator using the following scale: Excellent: complete control of asthma; Good: marked improvement of asthma; Moderate: discernible, but limited improvement in asthma; Poor: no appreciable change in asthma; Worsening of asthma
Time Frame: 20 Weeks
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Omalizumab + Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 76 | 37
Participants
  Excellent | 22 | 2
  Good | 35 | 4
  Moderate | 13 | 11
  Poor | 6 | 18
  Worsening | 0 | 2

10. Secondary Outcome: Patient's Global Assessment of Treatment Effectiveness
Description: At the end of Week 20, a global evaluation of the treatment effectiveness was performed by the patient using the following scale:
  Excellent: complete control of asthma; Good: marked improvement of asthma; Moderate: discernible, but limited improvement in asthma; Poor: no appreciable change in asthma; Worsening of asthma
Time Frame: 20 Weeks
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Omalizumab + Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 76 | 37
Participants
  Excellent | 33 | 3
  Good | 30 | 13
  Moderate | 10 | 10
  Poor | 3 | 9
  Worsening | 0 | 2

ADVERSE EVENTS:
Arm/Group | Omalizumab + Conventional Therapy | Conventional Therapy
Serious Adverse Events (participants affected / at risk) | 3/78 | 0/38
Other Adverse Events (participants affected / at risk) | 42/78 | 16/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab + Conventional Therapy (N=78) | Conventional Therapy (N=38)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab + Conventional Therapy (N=78) | Conventional Therapy (N=38)
Pyrexia (General disorders) | 4 | 0
Joint sprain (Injury, poisoning and procedural complications) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 1
Headache (Nervous system disorders) | 16 | 4
Anxiety (Psychiatric disorders) | 4 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.